CLINICAL TRIAL: NCT03814681
Title: Postoperative Outcomes Within/Without an Enhanced Recovery After Surgery Protocol in Colorectal Surgery Across Europe
Brief Title: Postopoperarive Outcomes After Colorectal Surgery in Europe (euroPOWER)
Acronym: EuroPOWER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Grupo Español de Rehabilitación Multimodal (Other)
Collaborators: GRACE Group (Other); REDGERM (Unknown)
Responsible Party: Sponsor
Other Study IDs: EuroPOWER
Record Dates: First submitted 2019-01-20; First posted 2019-01-24 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Perioperative Care; Colorectal Surgery; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Colorectal Surgery — elective Colorectal Surgery

SUMMARY:
Methods

30 days European Multicentre observational cohort study of postoperative complications following elective colorectal surgery within any compliance of an ERAS protocol (including patients with 0 compliance) in a participating hospital during the 30-day cohort period with a planned overnight stay.

Research sites

Hospitals across Europe with an elective colorrectal surgical service

Objective

To provide detailed data describing post-operative complications and associated mortality To provide detailed data describing adherence to ERAS protocol and its association to morbidity and length of stay.

To provide detailed information on the influence of the volume of patients undergoing surgery on each center and postoperative complications censured at 30 days after surgery.

Inclusion criteria All adult patients (aged ≥18 years) undergoing elective colorectal surgery during the 30-day study period.

Statistical analysis Number of patients: All eligible patients undergoing elective colorectal surgery during the study month in European participating hospitals.

Univariate analysis will be used to test factors (patient, surgical, and ERAS related) associated with surgical complications, length of stay (LOS) and in-hospital death. Single and multi-level logistic regression models will be constructed to identify factors independently associated with these outcomes and to adjust for differences in confounding factors. A stepwise approach will be used to enter new terms. A single final analysis is planned at the end of the study.

Summary statistics with post hoc Bonferroni corrections will be used to assess possible dose- response dependence in percentage of patients with postoperative complications and LOS.

DETAILED DESCRIPTION:
The results of this study will allow to identify, on the one hand, the type of patients presenting postoperative complications and, on the other hand, to identify those items of the ERAS protocols that are independently associated with a reduction in postoperative complications and hospital stay, which will allow to focus the perioperative efforts in those items that actually improve the postoperative outcomes.

* Aim 1 will establish the number of patients developing predefined postoperative complications within 30 days of surgery in adult patients undergoing elective colorectal surgery with any compliance of an ERAS protocol (including patients with 0 compliance). This will allow us to determine the actual impact of these protocols.
* Aim 2 will allow us to know the type of predefined complication presented by the patients included in the ERAS protocols and in patients undergoing colorectal surgery; This will allow, on the one hand, to have a starting point for future clinical trials, and, on the other hand, to focus efforts to avoid these complications.
* Aim 3 will allow us to identify those perioperative items of ERAS protocols that are actually associated with a decrease in postoperative complications.

The proposed study will establish a real view of the number of patients presenting postoperative complications that will overcome the limitations of available retrospective studies and provide greater insight into the items of the protocols that are associated with decreased complications; on the other hand, our hypothesis is that the number of patients who develop predefined postoperative complications within 30 days of surgery decreases as there is greater compliance with the predefined ERAS protocol items

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (aged ≥18 years) undergoing primary elective colorectal surgery and by any approach (Includes surgery with laparoscopic, assisted laparoscopic approach or open approach) in a participating hospital during the 30-day cohort period with a planned overnight stay.

Exclusion Criteria:

* Patients submitted for emergency surgery

  * Patients with complex cancer who required resection of organs other than bowel. (i.e. kidney, gastric resection, ovarian)• Patients treated with endoscopic techniques using the hybrid TaTME technique (Transanal Total Mesorectal Excision)
  * Bowel transit reconstruction surgery
  * Patients who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients (aged ≥18 years) undergoing primary elective colorectal surgery
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
Predefined mild-moderate-severe postoperative complications | 30 days after surgery
  Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine were published by the EPCO definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome mesures. infectious complications, cardiovascular complications and other types of complications. Each complication will be graded as mild, moderate or severe.

SECONDARY OUTCOMES:
In-hospital all-cause mortality | 30 days after surgery
  The number and percentage of deaths within 30 days of surgery will be reported for each surgical category
Compliance with ERAS items | 30 days after surgery
  Overall compliance will be calculated as the average of all pre- and intraoperative ERAS adapted elements, as specified in the ERAS society colon and rectal guidelines ERAS patients' guideline compliance will be categorised into quartiles
Duration of hospital stay | 30 days after surgery
  The median hospital length of stay (LOS) following the start of surgery, overall, by survival status and by complication status will be reported. Post-operative LOS is the duration in days from the date of the end of surgery to the date of discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Ripollés-Melchor, MD, Study Chair — Infanta Leonor University Hospital, Madrid, Spain; Rupert Pearse, Prof, Study Chair — Queen Mary University London, London, UK; José M Ramírez Rodríguez, Prof, Study Chair — Lozano Blesa University Hospital, Zaragoza, Spain; Samir Jaber, Prof, Study Chair — Hospitalier Universitaire de Montpellier, France; Karim Slim, Prof, Study Chair — Président de GRACE; César Aldecoa, Prof, Study Chair — Río Hortega University Hospital, Valladolid, Spain; Nader Francis, Prof, Study Chair — Yeovil District Hospital NHS Foundation Trust; Ane Abad-Motos, MD, Study Chair — Infanta Leonor University Hospital, Madrid, Spain
Locations (1):
- Hospital Universitario Infanta Leonor, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alves A, Panis Y, Mathieu P, Mantion G, Kwiatkowski F, Slim K; Association Francaise de Chirurgie. Postoperative mortality and morbidity in French patients undergoing colorectal surgery: results of a prospective multicenter study. Arch Surg. 2005 Mar;140(3):278-83, discussion 284. doi: 10.1001/archsurg.140.3.278. PMID 15781793
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, Macfie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):259-84. doi: 10.1007/s00268-012-1772-0. No abstract available. PMID 23052794
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT03814681/Prot_SAP_000.pdf